CLINICAL TRIAL: NCT05433207
Title: EDIROL Drug Intensive Monitoring: Post-Marketing Drug Intensive Monitoring Surveillance of EDIROL in Patients With Postmenopausal Osteoporosis
Brief Title: Post-Marketing Drug Intensive Monitoring Surveillance of EDIROL in Patients With Postmenopausal Osteoporosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: EDR2201CN
Record Dates: First submitted 2022-06-08; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Drug: Eldecalcitol soft capsules — 0.75 μg orally once a day during the intensive monitoring period. (The dose can be appropriately reduced to 0.5 μg according to symptoms, once a day.)

SUMMARY:
This is a post-marketing drug intensive monitoring surveillance with an observational, non-interventional design. The objectives are to compare the incidence of hypercalcemia in patients with and without calcium intake (including dietary supplements, excepting calcium from meals), and to monitor the type, incidence, severity, and relevance of other adverse drug reactions,including urolithiasis.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal osteoporosis patients who signed the informed consent form and are expected to receive Edirol during the intensive monitoring period.

  * Patients with postmenopausal osteoporosis
  * Patients who signed the informed consent form
  * Patients who are expected to receive Edirol during planned enrollment period

Exclusion Criteria:

* Exclude if any of the following:

  * Men
  * No osteoporosis
  * Other osteoporosis (not postmenopausal)
* Started Edirol before ICF signature
* Did not sign ICF

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Postmenopausal osteoporosis patients who signed the informed consent form and are expected to receive Edirol during the intensive monitoring period.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
the rates of hypercalcemia and 95% confidence intervals for patients with and without calcium preparation intake | one year from Edirol dosing date
the odds ratios of hypercalcemia and 95% confidence intervals for patients with and without calcium preparation intake | one year from Edirol dosing date
the proportion of each type of adverse drug reactions (including hypercalcemia, urolithiasis, etc.) | through study completion, up to one year
the incidence of adverse drug reactions (including hypercalcemia, urolithiasis, etc.) | through study completion, up to one year
the severity of adverse drug reactions (including hypercalcemia, urolithiasis, etc.) | through study completion, up to one year

CONTACTS AND LOCATIONS:
Overall Officials: Weibo Xia, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided